CLINICAL TRIAL: NCT06188338
Title: Clinical Study on 56-Day Continuous Improvement of 1064nm Fractional Picosecond Laser Treatment With Formulations of A Proprietary Anti-aging Complex Composition
Brief Title: A 56-day Clinical Study on Facial Skin Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Botanee Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C23021036
Record Dates: First submitted 2023-12-06; First posted 2024-01-03 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2023-12

CONDITIONS: Skin Manifestations; Wrinkle; Photoaging
MeSH Terms: conditions — Skin Manifestations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formulation containing MLYAAT-1002® Composition (Active Comparator): After the 1064nm fractional picosecond laser treatment, daily use of the formulation for 56 days: apply one pump of the formulation to the treated side of the face in the morning and evening, respectively.
  Interventions: Combination Product: Fractional picosecond laser treatment followed by daily use of formulations containing MLYAAT-1002®.
- Blank formulation without MLYAAT-1002® Composition (Placebo Comparator): After the 1064nm fractional picosecond laser treatment, daily use of the blank formulation for 56 days: apply one pump of the blank formulation to the control side of the face in the morning and evening, respectively.
  Interventions: Combination Product: Fractional picosecond laser treatment followed by daily use of formulations without MLYAAT-1002®

INTERVENTIONS:
Combination Product: Fractional picosecond laser treatment followed by daily use of formulations containing MLYAAT-1002®. — Each subject will receive a single treatment of the fractional picosecond laser, followed by the first application of the active comparator on the randomly assigned side of the split-face (the treatment side) on the same day, and sequently, will apply the active comparator to this side twice a day for 56 days.
  Arms: Formulation containing MLYAAT-1002® Composition
Combination Product: Fractional picosecond laser treatment followed by daily use of formulations without MLYAAT-1002® — Each subject will receive a single treatment of the fractional picosecond laser, followed by the first application of the placebo comparator on the randomly assigned side of the split-face (the control side) on the same day, and sequently, will apply the placebo comparator to this side twice a day for 56 days.
  Arms: Blank formulation without MLYAAT-1002® Composition

SUMMARY:
This clinical trial aims to learn about the efficacy of MLYAAT-1002® (a proprietary anti-aging complex, MLYAAT is short for "multi-layer anti-ageing technology" ) in female subjects who have newly received the rejuvenation treatment by comparing visual clinical scores, skin attributes measurement and image analysis.

DETAILED DESCRIPTION:
The main expectations are:

* After the 8-week continuous use of the test formulations with MLYAAT-1002® on one split-face side, the clinical manifestations and scores of photoaging improve compared to those of the control side using the placebo formulations.
* After the 8-week continuous use of the test formulations with MLYAAT-1002®, indicators of skin tone, individual type angle (ITA), CIELAB color space, pores and wrinkles improve compared to those of the control side using the placebo formulations.

ELIGIBILITY:
Inclusion Criteria:

* self-reported facial aging problems such as roughness, fine lines, and dull skin
* no symptoms of itching, tingling, or burning on the face
* no symptoms of facial flushing, erythema, papules, desquamation, or spot haemorrhage as evaluated by a dermatologist
* photodamage scores above 2 (evaluated by a dermatologist)
* compliance with split-face use of the assigned formulations for 56 days
* no antibiotics remedy in the past three months
* regular use of sunscreen products at least five times a week
* no plans to leave Shanghai during the period of the trial
* compliance with no use of any cosmetics that may bias the study results during the period of the trial
* written informed consent and portrait right consent were obtained from all participants before study entry

Exclusion Criteria:

* female subjects who are pregnant, lactating or planning to become pregnant
* history of alcoholism
* history of allergies
* subjects who have received medical rejuvenation treatment within the past one year
* being a participant in any other clinical trial within the past one month
* subjects who are suffering from facial skin diseases (melasma, acne, and herpes simplex, etc.)
* subjects with scar constitution or that predispose to Koebner's phenomenon (such as vitiligo and lichen planus, etc.)
* subjects who had skin diseases (such as psoriasis, eczema, and skin cancer, etc.)
* taken/injected anti-allergy medication in the past one month
* subjects who had a high fever in the past 2 weeks
* received anticancer chemotherapy or immunotherapy in the past 6 months
* anyone that the investigator thinks of not eligible.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-18 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
changes in skin manifestations of photodamage (global score) | Day 0, Day 15, Day 29, Day 57
  Scoring by two independent dermatologists, a global score of facial skin on a 5-point scale (0-4) will be recorded, i.e., lower scores meaning a better outcome.
changes in skin manifestations of photodamage (tactile skin roughness) | Day 0, Day 15, Day 29, Day 57
  Scoring by two independent dermatologists, a roughness score of facial skin on a 5-point scale (0-4) will be recorded, i.e., lower scores meaning a better outcome.
changes in skin manifestations of photodamage (fine lines) | Day 0, Day 15, Day 29, Day 57
  Scoring by two independent dermatologists, a fine-line score of facial skin on a 5-point scale (0-4) will be recorded, i.e., lower scores meaning a better outcome.
changes in skin manifestations of photodamage (coarse wrinkles) | Day 0, Day 15, Day 29, Day 57
  Scoring by two independent dermatologists, a coarse-wrinkle score of facial skin on a 5-point scale (0-4) will be recorded, i.e., lower scores meaning a better outcome.
changes in skin manifestations of photodamage (mottled pigmentation) | Day 0, Day 15, Day 29, Day 57
  Scoring by two independent dermatologists, a pigmentation score of facial skin on a 5-point scale (0-4) will be recorded, i.e., lower scores meaning a better outcome.
changes in skin manifestations of photodamage (erythema) | Day 0, Day 15, Day 29, Day 57
  Scoring by two independent dermatologists, an erythema score of facial skin on a 5-point scale (0-4) will be recorded, i.e., lower scores meaning a better outcome.
changes in skin manifestations of photodamage (dull skin) | Day 0, Day 15, Day 29, Day 57
  Scoring by two independent dermatologists, a dull-skin score of facial skin on a 5-point scale (0-4) will be recorded, i.e., lower scores meaning a better outcome.
changes in skin manifestations of photodamage (telangiectasia) | Day 0, Day 15, Day 29, Day 57
  Scoring by two independent dermatologists, a telangiectasia score of facial skin on a 5-point scale (0-4) will be recorded, i.e., lower scores meaning a better outcome.

SECONDARY OUTCOMES:
changes in skin surface hydration(a.u.) of facial skin | Day 0, Day 3, Day 5, Day 8, Day15, Day 29, Day 57
  measuring hydration of the stratum corneum by Corneometer® MPA580 (Courage&Khazaka#Germany)
changes in transepidermal water loss (TEWL#in g/m2/h) of facial skin | Day 0, Day 3, Day 5, Day 8, Day15, Day 29, Day 57
  measuring the loss of water that passes from inside a body through the epidermis to the surrounding atmosphere by Tewameter® MPA580 (Courage&Khazaka#Germany)
changes in index of erythema of facial skin | Day 0, Day 3, Day 5, Day 8, Day15, Day 29, Day 57
  measuring erythema by Mexameter MX18(Courage&Khazaka, Germany)
changes in index of melanin of facial skin | Day 0, Day 3, Day 5, Day 8, Day15, Day 29, Day 57
  measuring melanin by Mexameter MX18(Courage&Khazaka, Germany)
changes in individual typology angle (ITA°) of facial skin | Day 0, Day 1, Day 3, Day 5, Day 8, Day15, Day 29, Day 57
  capturing facial images by VISIA-7 (CANFIELD, America) and calculating the ITA
changes in the percentage of facial skin pore area | Day 0, Day 1, Day 3, Day 5, Day 8, Day15, Day 29, Day 57
  capturing facial images by VISIA-7 (CANFIELD, America) and calculating the percentage of pore area
changes in the characteristics of facial wrinkles （depth) | Day 0, Day 1, Day 3, Day 5, Day 8, Day15, Day 29, Day 57
  capturing facial images by VISIA-7 (CANFIELD, America), and recording the depth of wrinkles at the specific face region
changes in the characteristics of facial wrinkles | Day 0, Day 1, Day 3, Day 5, Day 8, Day15, Day 29, Day 57
  capturing facial images by VISIA-7 (CANFIELD, America), and recording the area of wrinkles at the specific face region
changes in the characteristics of crow's feet | Day 0, Day 29, Day 57
  capturing facial images by Primos (CANFIELD, America) and calculating the area of crow's feet at the specific face region
safety and tolerability | Day 0, Day 1, Day 3, Day 5, Day 8, Day15, Day 29, Day 57
  Any adverse effects (e.g., erythema, flush, stinging, pruritus, and spot hemorrhage, desquamation) on both sides of face will be recorded at each visit by two independent dermatologists. The severity of the observed effect will be scored on a 5-point scale (0-4) , i.e., higher scores meaning a more severe level .
self-assessment by participants | Day 0, Day 1, Day 3, Day 5, Day 8, Day15, Day 29, Day 57
  All the particpants will be asked to report any discomfort (e.g., stinging, pruritus, burning sensation) in their faces at each visit. The severity of the reported discomfort will be scored on a 5-point scale (0-4) , i.e., higher scores meaning a more severe level.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Shuxian, Dr, Principal Investigator — Shanghai Yaokang Clinic
Locations (1):
- Shanghai China-norm Quality Technical Service Co ，Ltd, Shanghai, Shanghai Municipality, China